CLINICAL TRIAL: NCT04458181
Title: Journaling and Addiction Recovery: Piloting "Positive Recovery Journaling"
Acronym: PPJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004619-2
Record Dates: First submitted 2020-05-21; First posted 2020-07-07 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants in this group will complete the intervention, Positive Peer Journaling (PPJ), while also continuing to attend intensive outpatient treatment for addiction.
  Interventions: Behavioral: Positive Peer Journaling (PPJ)
- Control Group (No Intervention): There will be no intervention for those randomized to the control group. However, they will complete assessment instruments throughout the study period while also continuing to attend intensive outpatient treatment for addiction.

INTERVENTIONS:
Behavioral: Positive Peer Journaling (PPJ) — PPJ is a journaling practice to support addiction recovery. PPJ encourages past 24 hour review and upcoming 24 hour planning to improve subjective wellbeing in recovery and reduce relapse. PPJ uses journals with column headings under which individuals make bullet-pointed lists. On the left hand page, past 24 hours is recalled, itemizing "good" and "bad" things that happened and things for which one is grateful. Good wishes for others are also expressed on this page. On the right hand page, values-based activities for the upcoming 24 hours are planned via headings representing valued life domains such as "recovery," "work/school," "spirituality," "home and household," and "health."
  Arms: Treatment Group

SUMMARY:
The main objective of this study is to pilot test the Positive Peer Journaling (PPJ) [later renamed "Positive Recovery Journaling" (PRJ)] intervention and its feasibility and acceptability. A second objective is to compare individuals assigned to PPJ to individuals in a treatment as usual control group.

DETAILED DESCRIPTION:
Many spiritual and religious traditions involve the practice of personal inventory and self-examination. These practices involve conducting a review of the day, spirituality, gratitude, and striving for self-knowledge and self-improvement. The 10th step of Alcoholics Anonymous (AA) recommends that members conduct such a daily inventory. While this practice may benefit AA members, not everyone seeking addiction recovery joins AA. Even for those who do, it can take time to reach step 10 and begin deriving benefits from it. The study PI, Dr. Amy Krentzman, developed Positive Recovery Journaling (PRJ, formerly "positive peer journaling") as a simple 10-minute daily practice which reviews the past 24 hours on the left side of a journal page and plans the upcoming 24 hours on the right side of a journal page. The prompts for the left and right sides of the PRJ page are based on principles from positive psychology and behavioral activation.

The main objective of this study is to pilot test the PRJ intervention and to examine the feasibility, acceptability, and logistics of treatment delivery.

A second objective is to observe whether PRJ is associated with improvement in satisfaction with life, happiness with recovery, and commitment to sobriety

ELIGIBILITY:
Inclusion Criteria:

* meet DSM-V criteria for past-year Substance Use Disorder as primary or secondary diagnosis,
* English literacy sufficient to make short written lists needed to complete PPJ and homework assessments,
* minimum 2 weeks sustained abstinence,
* completed first 2 weeks of treatment at Nuway (approximately 2 weeks), an intensive outpatient substance use disorder treatment program and the recruitment site,
* agree to be audio recorded or transcription recorded in group meetings and in individual meetings with research staff,
* currently are clients in the Nuway outpatient program,
* participants must be English speaking and literacy must be strong enough to write short lists and to understand the questions asked in the questionnaires,
* participants must have an electronic device that connects to the internet and internet connection for online delivery of intervention during COVID-19.

Exclusion Criteria:

* presence of a psychotic disorder, psychiatric condition (e.g., suicidal ideation), or cognitive impairment (e.g., severe dementia, traumatic brain injury) limiting ability to give consent and/or participate in the study;
* severe psychiatric illness (current schizophrenia, major depression with suicidal ideation);
* personality disorders that would interfere with satisfactory participation in or completion of the study protocol,
* inability to give informed, voluntary consent to participate,
* lack of sufficient English literacy to participate, defined as inability to make a list of 5 things they did yesterday and inability to understand questionnaire items,
* any impairment, activity, or situation that in the judgement of the research staff would prevent satisfactory participation in or completion of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Krentzman, MSW, PhD, Principal Investigator — University of Minenesota
Locations (1):
- NUWAY, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 42 | 39
Completed | 22 | 28
Not Completed | 20 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.7) | 39.4 (10.4) | 39 (11)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 18 | 19 | 37
  Female | 24 | 19 | 43
  Non Binary | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 28 | 32 | 60
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Life at Baseline
Description: Score on the "Satisfaction with Life" scale. This scale has 5 items assessed on a 7 point Likert-type response format. Scores range from 5 to 35 with higher scores representing higher satisfaction with life.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 42 | 39
units on a scale | 17.8 (6.6) | 17.2 (6.4)

2. Primary Outcome: Satisfaction With Life at 2 Weeks
Description: as for outcome 1
Time Frame: 2 weeks (after Phase 1, the group phase)
Population: The "Overall Number of Participants Analyzed" reported here represents the study census for this outcome at 2 weeks. In the study flow section of this report, the values reported under "completed" represent the study census at 8 weeks. That is why the values reported here and the values reported in the study flow under "completed" do not match.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 35
units on a scale | 20.5 (6.8) | 18.6 (7.8)

3. Primary Outcome: Satisfaction With Life at 4 Weeks
Description: as for outcome 1
Time Frame: 4 weeks (after Phase 2, the independent practice phase)
Population: The "Overall Number of Participants Analyzed" reported here represents the study census for this outcome at 4 weeks. In the study flow section of this report, the values reported under "completed" represent the study census at 8 weeks. That is why the values reported here and the values reported in the study flow under "completed" do not match.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 24 | 31
units on a scale | 19.4 (7.5) | 18.8 (7.9)

4. Primary Outcome: Satisfaction With Life at 8 Weeks
Description: as for outcome 1
Time Frame: 8 weeks (the 1-month post-intervention)
Population: The "Overall Number of Participants Analyzed" reported here represents the study census for this outcome at 8 weeks. These values match the values reported as "completed" in the study flow section of this report.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 22 | 28
units on a scale | 21 (7.4) | 21.2 (7.9)

5. Primary Outcome: Happiness With Recovery at Baseline
Description: Score on a single item, "In general, I am happy with my recovery." This item uses an 11 point scale ranging from 0 to 10. Higher scores represent higher happiness with recovery.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
units on a scale | 8.1 (1.9) | 8.4 (1.8)

6. Primary Outcome: Happiness With Recovery at 2 Weeks
Description: as for outcome 5
Time Frame: 2 weeks (after Phase 1, the group phase)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 35
units on a scale | 8.3 (1.8) | 8.6 (1.9)

7. Primary Outcome: Happiness With Recovery at 4 Weeks
Description: as for outcome 5
Time Frame: 4 weeks (after Phase 2, the independent practice phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 24 | 31
units on a scale | 8.4 (2.2) | 8.4 (1.9)

8. Primary Outcome: Happiness With Recovery at 8 Weeks
Description: as for outcome 5
Time Frame: 8 weeks (the 1-month post intervention)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 22 | 28
units on a scale | 8.2 (2) | 8.3 (2.4)

9. Primary Outcome: Commitment to Sobriety at Baseline
Description: Score on a single item, "I am willing to do whatever it takes to recover from my addiction." This item uses an 11 point scale ranging from 0-10. Higher scores represent greater commitment to sobriety.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 42 | 38
units on a scale | 8.6 (1.8) | 9.2 (1.4)

10. Primary Outcome: Commitment to Sobriety at 2 Weeks
Description: as for outcome 9
Time Frame: 2 weeks (after Phase 1, the group phase)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 26 | 35
units on a scale | 8.8 (1.5) | 9.1 (1.7)

11. Primary Outcome: Commitment to Sobriety at 4 Weeks
Description: as for outcome 9
Time Frame: 4 weeks (after Phase 2, the independent practice phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 24 | 31
units on a scale | 8.8 (1.5) | 8.9 (1.8)

12. Primary Outcome: Commitment to Sobriety at 8 Weeks
Description: as for outcome 9
Time Frame: 8 weeks (the 1-month post intervention)
Population: The "Overall Number of Participants Analyzed" reported here represents the study census for this outcome at 8 weeks. These values match those reported as "completed" in the the study flow section of this report.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 22 | 28
units on a scale | 8.5 (2.5) | 8.6 (2.1)

ADVERSE EVENTS:
Time Frame: From baseline screening through 8 week assessment (approximately 8 weeks).
Description: The study team monitored all participant communication including but not limited to Zoom screenings and group sessions, as well as written communication in the PRJ journals, for information of concern to health or wellbeing.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/39
Other Adverse Events (participants affected / at risk) | 0/42 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT04458181/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT04458181/ICF_001.pdf